CLINICAL TRIAL: NCT06376669
Title: Prospective Phase II Study of Stereotactic Body Proton Therapy for Treatment of PrimAry Renal Cell Carcinoma (SPARE)
Brief Title: Stereotactic Body Proton Therapy for Treatment of Primary Renal Cell Carcinoma
Acronym: SPARE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Robert L. Sloan Fund for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2421; IRB00427823 (Other: JHM IRB)
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Renal Cell Carcinoma
Keywords: Stereotactic Body Radiation Therapy; SBRT; RCC
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proton Stereotactic Body Radiation Therapy (SBRT) (Experimental): The SBRT group is the single arm of this study.
  Interventions: Radiation: Proton Stereotactic Body Radiation therapy (SBRT)

INTERVENTIONS:
Radiation: Proton Stereotactic Body Radiation therapy (SBRT) — Radiation therapy will consist of 3-5 treatments over 1.5 - 2 weeks

SUMMARY:
This study examines the impact of proton based stereotactic radiation therapy (SBRT) on kidney function as well as other oncologic outcomes including local control, locoregional and systemic failure, progression free and overall survival.

DETAILED DESCRIPTION:
The incidence of kidney cancer diagnosis has been increasing over the last years. Surgical resection represents the mainstay treatment. However, many patients are deemed unfit for surgery due to medical comorbidities or technical limitations. There are non-surgical options including active surveillance, cryotherapy, microwave ablation, radiofrequency and stereotactic radiation therapy (SBRT). SBRT using conventional x-rays has recently been shown to improve outcomes for patients with primary renal cell carcinoma (RCC) in terms of local control and toxicity. However, this treatment was associated with a significant decline in kidney function that necessitates additional intervention including dialysis in some patients. Proton therapy represents an emerging technique with unique properties that allow the bulk of the proton cancer fighting energy to be released at the tumor (Bragg peak) while sparing nearby healthy tissues and organs, particularly the remaining healthy kidney, ipsilateral kidney, bowels, spine and liver. With this technology, both kidneys, the remaining ipsilateral and contralateral, could be spared and thus less damage is expected. This study aims to study the impact of proton based SBRT on the kidney function.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Biopsy proven renal cell carcinoma.
3. No clinical or radiographic evidence of metastatic disease.
4. Not a candidate for surgical treatment or local ablative procedures.
5. Subjects are able to undergo either an MRI or administration of contrast agent for CT.

Exclusion Criteria:

1. Prior history of radiation treatment with overlapping fields.
2. Patients with proven metastatic disease.
3. Female subjects who are pregnant or planning to become pregnant during the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Change in kidney function after PROTON-BASED SBRT treatment as assessed by serum creatine levels | Baseline and every 3-6 months up to 2 years post treatment
  Change in serum creatine levels from Baseline visit.
Change in kidney function after PROTON-BASED SBRT treatment as assessed by estimated glomerular rate (eGFR) values | Baseline and every 3-6 months up to 2 years post treatment
  Change in eGFR values from Baseline visit.

SECONDARY OUTCOMES:
Number of PROTON-BASED SBRT treatment Adverse Events | 24 months post treatment
  Adverse events associated with PROTON-BASED SBRT treatment.
Local progression of disease after PROTON-BASED SBRT treatment as assessed by size or appearance of lesions | Baseline and every 3-6 months up to 2 years post treatment
  Local progression is defined as an increased size of the primary lesion or appearance of a new lesion in the kidney (within the radiation field).
Systemic progression of disease after PROTON-BASED SBRT treatment as assessed by appearance of lesions | Baseline and every 3-6 months up to 2 years post treatment
  Systemic progression is defined as appearance of new lesions outside the radiation field (away from the primary tumor).
Time to locoregional progression | Baseline and every 3-6 months up to 2 years post treatment
  Time to locoregional progression is defined as time from the date of first SBRT PROTON-BASED SBRT fraction to date of locoregional progression, according to RECIST v1.1 criteria.
Overall survival | 24 months post treatment
  Overall survival (OS) is defined as the duration of time from start of treatment to the time of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Shaaban, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Sibley Memorial Hospital, Washington D.C., District of Columbia, United States